CLINICAL TRIAL: NCT05629325
Title: The Effect of Oral Buspirone Hydrochloride on Esophageal Motility, Bolus Transit and Symptoms of Dysphagia, in Patients With Poor Esophageal Motility: A Randomized, Double-blind, Placebo Controlled, Cross-over Trial With HRiM
Brief Title: Buspirone for Weak or Absent Esophageal Peristalsis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S62876
Record Dates: First submitted 2022-11-08; First posted 2022-11-29 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Dysphagia, Esophageal
MeSH Terms: conditions — Deglutition Disorders | interventions — Buspirone

STUDY DESIGN:
Intervention Model Description: Patients with IEM or absent contractility and symptoms of dysphagia will participate in this study. They will be randomized on a 1:1 basis: Patients will be randomized to take buspirone for 4 weeks or placebo for 4 weeks. After a 2-week washout period the randomized groups will cross over into the alternate treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A randomization list will be prepared by the laboratorium Wolfs (Zwijndrecht, Belgium) and the trial medication will be labeled by the laboratorium Wolfs based on the randomization list. The randomization list is prepared separately from study investigators or coordinators. The participant, investigator and study team are blinded to the allocated treatment arm in both intervention periods (buspirone/placebo). Each study patient will be assigned a subsequent randomization number. If a medical emergency occurs and a decision about the subject's condition requires knowledge of the treatment assignment, the investigator will immediately notify the laboratorium Wolfs to break the blind for this individual subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Buspirone => Washout => Placebo (Experimental): Patients will take Buspirone hydrochloride 10mg oral once a day (in the evening) for 3 days, twice a day (morning and evening) for 4 days, three times a day for 2 weeks and 20mg oral three times a day for one week. Esophageal motility will be assessed with high resolution impedance manometry (HRiM) after 4 weeks of treatment. Patients will also report their perceived symptoms of dysphagia during the HRiM. A washout period of two weeks will take place. Afterwards, the second treatment period starts. Patients will take Placebo oral once a day (in the evening) for 3 days, twice a day (morning and evening) for 4 days, three times a day for 2 weeks and 20mg oral three times a day for one week. Esophageal motility will also be assessed with high resolution impedance manometry (HRiM) after 4 weeks of treatment. Patients will again report their perceived symptoms of dysphagia during the HRiM.
  Interventions: Drug: Buspirone Hydrochloride 10 MG; Drug: Placebo
- Placebo => Washout => Buspirone (Experimental): Patients will take Placebo oral once a day (in the evening) for 3 days, twice a day (morning and evening) for 4 days, three times a day for 2 weeks and 20mg oral three times a day for one week. Esophageal motility will be assessed with high resolution impedance manometry (HRiM) after 4 weeks of treatment. Patients will also report their perceived symptoms of dysphagia during the HRiM. A washout period of two weeks will take place. Afterwards, the second treatment period starts. Patients will take Buspirone hydrochloride oral once a day (in the evening) for 3 days, twice a day (morning and evening) for 4 days, three times a day for 2 weeks and 20mg oral three times a day for one week. Esophageal motility will also be assessed with high resolution impedance manometry (HRiM) after 4 weeks of treatment. Patients will again report their perceived symptoms of dysphagia during the HRiM.
  Interventions: Drug: Buspirone Hydrochloride 10 MG; Drug: Placebo

INTERVENTIONS:
Drug: Buspirone Hydrochloride 10 MG — 4 weeks of treatment with buspirone
  Other Names: Buspiron
Drug: Placebo — 4 weeks of treatment with placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, cross-over clinical trial of buspirone in patients with complaints of dysphagia due to poor esophageal motility. The goal of this clinical trial is to study the effect of buspirone on esophageal motility by performing high resolution impedance manometry (HRiM).

DETAILED DESCRIPTION:
Esophageal motility disorders can be characterized by poor esophageal motility with impaired clearance of the esophagus. Examples are Ineffective Esophageal Motility (IEM, >70% of the swallows are ineffective or ≥50% are failed) and Absent Contractility (100% failed peristalsis). Both might be the underlying cause for dysphagia.

Several studies have shown that poor esophageal motility can be manipulated by pharmacological means. Buspirone, a 5-HT1A agonist, is able to significantly increase distal esophageal wave amplitude and duration in healthy volunteers, suggesting it may be effective in IEM. At the moment, findings in patients with IEM are not consistent and depend on the dose and treatment duration.

This cross-over trial will examine the use of buspirone in patients with dysphagia, with the intent of using a higher dose. We will use impedance/manometry and pressure flow analysis to liquid, viscous and solid boluses to evaluate the symptomatic and manometric effect of buspirone.

ELIGIBILITY:
Inclusion Criteria:

Patients can participate in this study if:

1. A minimum of 18 years old;
2. Ineffective Esophageal Motility (IEM) or absent contractility, as determined on HRM in the last three months before inclusion in the study, using the Chicago classification v4.0 (1).

   IEM is defined as >70% ineffective or ≥50% failed swallows with a normal integrated relaxation pressure (IRP4). IEM includes a weak contraction (DCI ≥ 100 mmHg·s·cm and <450 mmHg·s·cm), failed peristalsis (DCI < 100 mmHg·s·cm), or fragmented peristalsis (a large break (>5 cm length) in the 20-mmHg isobaric contour with DCI > 450 mmHg·s·cm).

   Absent contractility is defined as 100% failed swallows (DCI < 100 mmHg·s·cm), with a normal IRP4.
3. Have completed a gastro-duodenoscopy, within 12 months, showing no anatomical abnormality of the stomach or esophagus, which can explain the patients' symptoms.
4. History of dysphagia for at least 2 months, at least twice per week in the last month.
5. Sexually active women of childbearing potential participating in the study must be using an appropriate form of contraception. Medically acceptable forms of contraception include oral contraceptives, injectable or implantable methods, intrauterine devices, or properly used barrier contraception. If the female patient has not been on oral, injectable, implantable or intrauterine contraception, a urinary pregnancy test will be performed prior to administration of Buspirone/Placebo.
6. Subjects must be capable of understanding and be willing to provide signed and dated written voluntary informed consent before any protocol-specific screening procedures are performed.

Exclusion Criteria:

Patients cannot participate in this study if:

1. Endoscopic signs of severe erosive esophagitis (grade C or D, Los Angeles classification) on endoscopy performed off PPI treatment in the 12 months prior to screening, or ≥ grade B when endoscopy is performed during PPI treatment.
2. Systemic diseases, known to affect esophageal motility (i.e. systemic sclerosis)
3. Surgery in the thorax or in the upper part of the abdomen (appendectomy and cholecystectomy are allowed).
4. Hiatal hernia ≥3 cm
5. QT c>450 ms.
6. Use of medication that effect cholinergic function such as anticholinergics, tricyclic antidepressants.
7. Concomitant promotility agents such as prucalopride or domperidone.
8. Concomitant use of more than one benzodiazepine.
9. Significant neurological, respiratory, hepatic, renal, hematological, cardiovascular, metabolic or gastrointestinal cerebrovascular disease as judged by the investigator.
10. Major psychiatric disorder.
11. Pregnancy or breastfeeding.
12. History of poor compliance.
13. History of/or current psychiatric illness that would interfere with ability to comply with protocol requirements or give informed consent.
14. History of alcohol or drug abuse that would interfere with ability to comply with protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
HRiM Manometric Features: DCI 5ml supine | During manometric assessment after 4 weeks of treatment
  Changes in distal contractile integral (DCI, in mmHg*s*cm) between buspirone and placebo. DCI is established on HRiM. As primary endpoint, we will focus on the values for DCI for the liquid bolus, 5 ml in supine position.

SECONDARY OUTCOMES:
Bolus passage score | During manometric assessment after 4 weeks of treatment
  Patients will evaluate the perception of each swallow during the manometric assessment via the following Likert score: 1-Normal, 2-Slow passage of bolus, 3-Stepwise passage, 4-Partial Blockage, 5-Complete Blockage.
HRiM Manometric Features: PCI | During manometric assessment after 4 weeks of treatment
  Pharyngeal Esophageal Contractile Integral (PCI es., mm.Hg.s.cm)
HRiM Manometric Features: DCI | During manometric assessment after 4 weeks of treatment
  Distal Esophageal Contractile Integral (DCI, mmHg.s.cm)
HRiM Manometric Features: Largest Break Size | During manometric assessment after 4 weeks of treatment
  Largest Break Size (cm)
HRiM Manometric Features: DL | During manometric assessment after 4 weeks of treatment
  Distal Latency (DL, s)
HRiM Manometric Features: IRP4s | During manometric assessment after 4 weeks of treatment
  Integrated Relaxation Pressure EGJ 4sec (IRP4s, mmHg)
HRiM Manometric Features: PFI | During manometric assessment after 4 weeks of treatment
  Pressure Flow Index (PFI, -)
HRiM Manometric Features: IR | During manometric assessment after 4 weeks of treatment
  Impedance Ratio (IR, -)
HRiM Manometric Features: DPA | During manometric assessment after 4 weeks of treatment
  Distension Pressure Accommodation Phase (DPA, mmHg)
HRiM Manometric Features: DPE | During manometric assessment after 4 weeks of treatment
  Distension Pressure Emptying Phase (DPE, mmHg)
HRiM Manometric Features: RP | During manometric assessment after 4 weeks of treatment
  Distal Ramp Pressure (RP, mmHg/s)
HRiM Manometric Features: CSI | During manometric assessment after 4 weeks of treatment
  Contractile Segment Impedance (CSI, Ohm)
HRiM Manometric Features: BPT | During manometric assessment after 4 weeks of treatment
  Bolus Presence Time (BPT, s)
HRiM Manometric Features: BFT | During manometric assessment after 4 weeks of treatment
  Bolus Flow Time (BFT, s)
HRiM Manometric Features: EGJ Rest.P | During manometric assessment after 4 weeks of treatment
  EGJ Resting Pressure (EGJ Rest.P, mmHg)
HRiM Manometric Features: EGJCI | During manometric assessment after 4 weeks of treatment
  EGJ Contractile Integral (EGJCI, mmHg.cm)
HRiM Manometric Features: LES-CD | During manometric assessment after 4 weeks of treatment
  Lower Esophageal Sphincter - Crural Diaphragm (LES-CD, mm)
Mayo Dysphagia Questionnaire | At baseline and after 4 weeks of treatment
  Symptom questionnaire
Overall Treatment Evaluation (OTE) | At baseline and after 4 weeks of treatment
  Symptoms questionnaire
Overall Symptom Severity (OSS) | At baseline and after 4 weeks of treatment
  Symptom questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No